CLINICAL TRIAL: NCT05814757
Title: A Randomized, Double-masked, Study to Evaluate the Efficacy and Safety of OTX-DED (Dexamethasone Intracanalicular Ophthalmic Insert) for the Short-term Treatment of the Symptoms of Dry Eye Disease (DED)
Brief Title: OTX-DED for the Short-term Treatment of the Symptoms of Dry Eye Disease (DED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-DED-2022-C01
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Syndromes; Eye Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases | interventions — Punctal Plugs

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Masked Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OTX-DED 0.3mg (Experimental)
  Interventions: Drug: OTX-DED
- Controlled Insertion utilizing Collagen Punctal Plug (Experimental)
  Interventions: Drug: Controlled Insertion
- Collagen Punctal Plug (Full Insertion) (Placebo Comparator)
  Interventions: Drug: Collagen Punctal Plug

INTERVENTIONS:
Drug: OTX-DED — 0.3mg dexamethasone ophthalmic insert
  Arms: OTX-DED 0.3mg
Drug: Controlled Insertion — Collagen Punctal Plug 0.2mm (Controlled Insertion)
  Arms: Controlled Insertion utilizing Collagen Punctal Plug
Drug: Collagen Punctal Plug — Collagen Punctal Plug 0.2mm (Full Insertion)
  Arms: Collagen Punctal Plug (Full Insertion)

SUMMARY:
To assess the efficacy and safety of OTX-DED for the short-term treatment of the symptoms of DED

DETAILED DESCRIPTION:
Randomized, double-masked, study to evaluate the efficacy and safety of OTX-DED (dexamethasone intracanalicular ophthalmic insert) for the short-term treatment of the symptoms of dry eye disease (DED). The subjects will be followed for approximately two months.

ELIGIBILITY:
Inclusion Criteria:

* VAS eye dryness severity score ≥ 35 and ≤ 90 at screening.
* Investigator assessment of bulbar conjunctival hyperemia grade ≥ 2 (CCLRU; 0 - 4 scale).
* Unanesthetized Schirmer of > 0 and ≤ 10 mm.
* Must not have used Artificial Tears during the Screening period.
* IOP in both eyes ≥ 5 mmHg and ≤21 mmHg.

Exclusion Criteria:

* Have worn contact lenses in the 4 weeks prior to the screening visit and/or are unwilling to discontinue use of contact lenses throughout the study period.
* Have a history of glaucoma or ocular hypertension or have a history of intraocular pressure (IOP) < 5 mmHg or > 24 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Severity of Eye Dryness Score (visual analogue scale (VAS)) | Change from baseline (CFB) at Day 15
  Visual Analogue Scale (0 mm - no discomfort to 100mm - maximal (the most) discomfort)

CONTACTS AND LOCATIONS:
Locations (1):
- Ocular Therapeutix, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No